CLINICAL TRIAL: NCT02051582
Title: Role of the Laser Pointer in Budgeting Fluoroscopy Time and Radiation Exposure
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 201300829
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgeons using fluoroscopy with laser pointer: Surgeons will attempt to obtain a "perfect" anterior-posterior (AP) and axillary views of a cadaver wrist using a mini-fluoroscopy unit equipped with a laser pointer.
  A "perfect" view is considered the ability to obtain perfect circle views through a cannulated mini acutrak screw that will have been placed into the cadaver prior to data collection.
  Surgeons will also be asked to wear three dosimeter badges: one on the collar, one on the waist, and a ring badge under a pair of regular sterile surgical gloves.
  Interventions: Procedure: Surgeons using fluoroscopy with laser pointer
- Surgeons using fluoroscopy without laser pointer: Surgeons will attempt to obtain a "perfect" anterior-posterior (AP) and axillary views of a cadaver wrist using a mini-fluoroscopy unit equipped without a laser pointer.
  A "perfect" view is considered the ability to obtain perfect circle views through a cannulated mini acutrak screw that will have been placed into the cadaver prior to data collection.
  Surgeons will also be asked to wear three dosimeter badges: one on the collar, one on the waist, and a ring badge under a pair of regular sterile surgical gloves.
  Interventions: Procedure: Surgeons using fluoroscopy without laser pointer

INTERVENTIONS:
Procedure: Surgeons using fluoroscopy with laser pointer — Surgeons will attempt to obtain a "perfect" anterior-posterior (AP) and axillary views of a cadaver wrist using a mini-fluoroscopy unit equipped with a laser pointer.
  A "perfect" view is considered the ability to obtain perfect circle views through a cannulated mini acutrak screw that will have been placed into the cadaver prior to data collection.
  Surgeons will also be asked to wear three dosimeter badges: one on the collar, one on the waist, and a ring badge under a pair of regular sterile surgical gloves.
  Groups: Surgeons using fluoroscopy with laser pointer
Procedure: Surgeons using fluoroscopy without laser pointer — Surgeons will attempt to obtain a "perfect" anterior-posterior (AP) and axillary views of a cadaver wrist using a mini-fluoroscopy unit equipped without a laser pointer.
  A "perfect" view is considered the ability to obtain perfect circle views through a cannulated mini acutrak screw that will have been placed into the cadaver prior to data collection.
  Surgeons will also be asked to wear three dosimeter badges: one on the collar, one on the waist, and a ring badge under a pair of regular sterile surgical gloves.
  Groups: Surgeons using fluoroscopy without laser pointer

SUMMARY:
Thirty (30) orthopaedic surgeons from the University of Florida Department of Orthopaedics and Rehabilitation will be recruited and enrolled in the study to determine whether having a laser pointed on a fluoroscopy machine can significantly decrease the amount of radiation exposure as measured while obtaining multiple views during surgery as well as decrease radiation exposure and time to accomplish the goals of surgery.

DETAILED DESCRIPTION:
The subject be asked to participate in one test session at the UF Psychomotor and Surgical Skills Lab located in the UF Orthopaedics & Sports Medicine Institute. During this test session the patient will be asked to wear a 0.5mm thick lead wrap-around apron and thyroid shield for maximal protection from radiation. The patient will also be asked to wear three dosimeter badges: one on the collar, one on the waist, and a ring badge under a pair of regular sterile surgical gloves.

The patient will attempt to obtain a "perfect" anterior-posterior (AP) and axillary views of a cadaver wrist using a mini-fluoroscopy unit equipped with a laser pointer.

A "perfect" view is considered the ability to obtain perfect circle views through a cannulated mini acutrak screw that will have been placed into the cadaver prior to data collection.

The patient will attempt to achieve the perfect views using the fluoroscopy unit with and without the laser pointer. The use of the laser pointer will be randomized by a randomization table that is prepared prior to testing. The patient's total fluoroscopy time and the number of shots you take for each task recorded. The investigators will also record the number of years training the patient has as an orthopaedic surgeon.

Female Participants: Because the radiation exposure from the fluoroscopy machine in this study might affect an unborn baby, the patient will not be allowed to participate in the study if they are pregnant. All women of childbearing potential must take a pregnancy test prior to participating in this study.

ELIGIBILITY:
Inclusion Criteria:

orthopaedic surgeons (Attendings, Fellows, and Residents) from the Department of Orthopaedics and Rehabilitation

Exclusion Criteria:

non-orthopaedic surgeons (Attendings, Fellows, and Residents) from the Department of Orthopaedics and Rehabilitation

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty (30) orthopaedic surgeons (Attendings, Fellows, and Residents) from the Department of Orthopaedics and Rehabilitation will be recruited and enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Total radiation exposure with laser pointer will be measured. | 1 hour
  All dosimeters will be read for total radiation exposure. Data analysis will include simple statistics to compare the total radiation exposure and number of shots taken per task using each of the fluoroscopy machines with laser pointer.
Total radiation exposure without laser pointer will be measured. | 1 hours
  All dosimeters will be read for total radiation exposure. Data analysis will include simple statistics to compare the total radiation exposure and number of shots taken per task using each of the fluoroscopy machines without laser pointer.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Matthias, M.D., Principal Investigator — University of Florida
Locations (1):
- UF and Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States